CLINICAL TRIAL: NCT03848325
Title: Impact of Poor Sleep on Inflammation and the Adenosine Signaling Pathway in HIV Infection
Brief Title: Poor Sleep and Inflammation in HIV-Infected Adults
Acronym: SASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanjay R Patel, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO17120573; R01HL142118 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: HIV-1-infection; Sleep Deprivation; Inflammation
Keywords: adenosine
MeSH Terms: conditions — Sleep Deprivation; Inflammation

STUDY DESIGN:
Intervention Model Description: All participants will undergo one night of normal sleep (Night 1) followed by a subsequent night (Night 2) of sleep deprivation. Outcomes will be assessed the morning (Day 1 and Day 2) after each condition.
Masking Description: Technicians processing biospecimens will be blinded to whether samples were collected on Day 1 or Day 2. Similarly, the assessor of brachial artery reactivity measurements will be blinded to whether ultrasound images were collected on Day 1 or Day 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep deprivation (Experimental): All subjects will be provided an 8 hour opportunity for sleep (Night 1) followed by outcome assessment the next morning (Day 1). They will then be kept awake the subsequent 24 hours including Night 2, followed by outcome assessment the following morning (Day 2).
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — Eight hour opportunity for sleep followed by 24 hours of sleep deprivation.

SUMMARY:
People living with HIV (PLWH) often have poor sleep, which may put them at a higher risk for many chronic diseases, including cardiovascular disease. One of the mechanisms by which this may occur is via chronic inflammation and endothelial dysfunction. Adenosine plays an important role in sleep homeostasis, with levels increasing in the CSF in response to sleep deprivation and falling with sleep. Peripherally, adenosine, via its signaling pathway, plays an important role in immunoregulation by suppressing the inflammatory response. PLWH, even on antiretroviral therapy, have suppressed peripheral adenosine levels which are predictive of adverse cardiovascular outcomes. The hypothesis underlying this study is that acute sleep deprivation in PLWH does not result in a compensatory increase in extracellular adenosine and its signaling peripherally, and this failure to appropriately compensate, leads to an increase in systemic inflammation and endothelial dysfunction.

DETAILED DESCRIPTION:
People living with HIV infection (PLWH) are known to be at higher risk of cardiovascular disease and also have a higher prevalence of poor sleep than people who do not have HIV infection. Understanding the underlying mechanisms for the elevated risk of cardiovascular disease in PLWH is important to developing novel strategies to mitigate this risk. Poor sleep has been postulated to mediate some of the elevated cardiovascular risk in PLWH given the high prevalence of poor sleep in PLWH and the epidemiologic association of poor sleep with adverse cardiovascular outcomes among people who do not have HIV infection. However, the mechanisms by which PLWH may be more sensitive to sleep loss from a cardiovascular standpoint are unclear. One potential explanation for any elevated sensitivity would be via alterations in the adenosine signaling pathway.

Changes in extracellular adenosine levels in the brain and central nervous system play an important homeostatic role in sleep-wake regulation. Sleep deprivation results in a rise in extracellular adenosine levels while sleep itself leads to a rapid decline in levels. Peripheral adenosine signaling is a central feature of immunoregulation, primarily through its effects on inflammatory cytokine expression and lymphocyte adenosine receptor expression. PLWH tend to have a suppressed level of peripheral adenosine signaling and this level of suppression predicts risk of cardiovascular disease. The purpose of this study is to explore the impact of acute sleep deprivation among PLWH on measures of inflammation and endothelial function and to assess the extent to which any changes may be explained by alterations in peripheral adenosine signaling.

The study will enroll 40 PLWH, age 18-75, who have been on ART for greater than 48 weeks. Screening with questionnaires, actigraphy and polysomnography will eliminate individuals with underlying chronic sleep abnormalities. A prior night of polysomnography in the sleep lab will also habituate subjects to sleeping while monitored in the sleep lab.

Participants will arrive in the sleep laboratory in the evening and be allowed to sleep for 8 hours timed to their usual sleep patterns. On waking, participants will provide a urine sample that will be assayed for adenosine and adenosine metabolites. Blood will be drawn to measure markers of inflammation as well as markers of activation of the peripheral adenosine signaling system. Endothelial function will be assessed using flow mediated dilation.

Participants will be kept awake for the subsequent 24 hours including the 8 hour normal sleep period. On the second morning, subjects will again provide urine and blood samples for the same bioassays described above and then undergo repeat assessment of endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* On continuous anti-retroviral therapy regimen for at least 48 weeks
* CD4+ cell count greater than or equal to 200 cells/mm^3

Exclusion Criteria:

* Irregular or insufficient habitual sleep patterns
* Severe advanced or delayed sleep phase
* Primary sleep disorder
* Autoimmune disorder
* Use of immunosuppressant medications
* Use of medications impacting adenosine pathway
* Heavy caffeine use
* Active alcohol or drug abuse
* Elevated risk of adverse health effects from sleep deprivation (e.g., bipolar disorder, epilepsy, or suicidal ideation in the past 6 months)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay R Patel, MD, Principal Investigator — University of Pittsburgh; Bernard J Macatangay, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep Repletion Followed by Sleep Deprivation: An 8 hour opportunity for sleep followed by outcome assessment the next morning and then 24 hour sleep deprivation followed by repeat outcome assessment.
Period: Overall Study
Arm/Group | Sleep Repletion Followed by Sleep Deprivation
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline (Sleep Repletion) Followed by Sleep Deprivation: An 8 hour opportunity for sleep followed by outcome assessment the next morning and then 24 hour sleep deprivation followed by repeat outcome assessment.
Arm/Group | Baseline (Sleep Repletion) Followed by Sleep Deprivation
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 10
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Soluble CD14
Description: Plasma concentration of soluble CD14
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation: An 8 hour opportunity for sleep followed by outcome assessment the next morning and then 24 hour sleep deprivation followed by repeat outcome assessment.
Arm/Group | Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation
Number analyzed (Participants) | 20
ng/mL
  Baseline (Sleep repletion) | 1290 (405)
  After sleep deprivation | 1196 (533)

2. Primary Outcome: Soluble CD163
Description: Plasma concentration of soluble CD163
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Population: All 20 participants who completed the protocol and whose blood sample met quality control for the assay performed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sleep Repletion Followed by Sleep Deprivation
Number analyzed (Participants) | 20
ng/mL
  Baseline (Sleep repletion): number analyzed (Participants) | 19
  Baseline (Sleep repletion) | 359 (231)
  After sleep deprivation: number analyzed (Participants) | 18
  After sleep deprivation | 384 (250)

3. Primary Outcome: IL6
Description: Plasma concentration of interleukin-6
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Population: All 20 participants who completed the protocol and whose blood sample met quality control for the assay performed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sleep Deprivation
Number analyzed (Participants) | 20
pg/mL
  Baseline (Sleep repletion): number analyzed (Participants) | 19
  Baseline (Sleep repletion) | 4.46 (2.06)
  After sleep deprivation: number analyzed (Participants) | 18
  After sleep deprivation | 4.27 (1.14)

4. Secondary Outcome: Flow Mediated Brachial Artery Dilation
Description: Percent change was calculated by measuring the brachial artery diameter at baseline and then the percent dilation from this baseline after release of occlusion at each time point.
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation
Number analyzed (Participants) | 20
% change
  Baseline (Sleep repletion) | 6.13 (2.68)
  After sleep deprivation | 4.42 (3.22)

5. Secondary Outcome: Monocyte Expression of IL6
Description: Percentage of circulating CD14+ peripheral blood mononuclear cells expressing interleukin-6
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Measure: Mean (Standard Deviation); unit: % cells
Arm/Group | Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation
Number analyzed (Participants) | 20
% cells
  Baseline (Sleep repletion) | 84.6 (13.6)
  After sleep deprivation | 89.1 (8.3)

6. Secondary Outcome: Monocyte Expression of TNF-alpha
Description: Percentage of circulating CD14+ peripheral blood mononuclear cells expressing tumor necrosis factor-alpha
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Measure: Mean (Standard Deviation); unit: % cells
Arm/Group | Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation
Number analyzed (Participants) | 20
% cells
  Baseline (Sleep repletion) | 52.0 (37.4)
  After sleep deprivation | 64.1 (32.4)

7. Secondary Outcome: CD4+ T-cell Expression of HLA-DR and CD38
Description: Percentage of CD3+ CD4+ T-lymphocytes co-expressing HLA-DR and CD38
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Measure: Mean (Standard Deviation); unit: % cells
Arm/Group | Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation
Number analyzed (Participants) | 20
% cells
  Baseline (Sleep repletion) | 8.14 (9.09)
  After sleep deprivation | 8.39 (9.01)

8. Secondary Outcome: CD8+ T-cell Expression of HLA-DR and CD38
Description: Percentage of CD3+ CD8+ T-lymphocytes co-expressing HLA-DR and CD38
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Measure: Mean (Standard Deviation); unit: % cells
Arm/Group | Baseline (Sleep Replete State) Followed by 24 Hours of Sleep Deprivation
Number analyzed (Participants) | 20
% cells
  Baseline (Sleep repletion) | 12.30 (10.74)
  After sleep deprivation | 13.17 (11.06)

9. Other Pre Specified Outcome: Plasma Adenosine
Description: Plasma adenosine concentration
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Plasma Inosine
Description: Plasma inosine concentration
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Urine 3'5'-cAMP
Description: Urine 3'5'-cyclic adenosine monophosphate concentration normalized to creatinine
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Reporting Status: Not Posted

12. Other Pre Specified Outcome: CD4+ T-cell Expression of CD39 and/or CD73
Description: Percentage of CD3+ CD4+ T-lymphocytes expressing CD39 and/or CD73
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Reporting Status: Not Posted

13. Other Pre Specified Outcome: CD8+ T-cell Expression of CD39 and/or CD73
Description: Percentage of CD3+ CD8+ T-lymphocytes expressing CD39 and/or CD73
Time Frame: Baseline sleep replete state and after 24 hours of sleep deprivation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Baseline (Sleep Repletion) Followed by Sleep Deprivation
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (Sleep Repletion) Followed by Sleep Deprivation (N=20)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) — Petechiae on arm from blood pressure cuff inflation for brachial artery reactivity testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT03848325/Prot_SAP_000.pdf